CLINICAL TRIAL: NCT07226531
Title: Retrospective Cohort Study to Assess Utilization and Effectiveness of Ritlecitinib in a Real-World Population With Severe Alopecia Areata in the United States
Brief Title: Utilization and Effectiveness of Ritlecitinib in a Real-World Population With Severe AA in the US
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7981121
Record Dates: First submitted 2025-09-22; First posted 2025-11-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alopecia areata (AA) patients treated with ritlecitinib
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — As provided in real-world practice

SUMMARY:
Alopecia areata (AA) is a chronic, relapsing T-cell mediated autoimmune disease characterized by nonscarring, typically patchy hair loss that affects people of all ages, races, and genders. In the United States (US), AA has an estimated point prevalence of 1.14% (Beningo et al., 2020). The three most common subtypes of AA are defined by the affected area:

* Patchy alopecia (PA), as seen in 90% of clinical diagnoses: hair loss occurring in one or more patches (ranging from coin-sized to large patches and even full scalp involvement) on the scalp or other parts of the body;
* Alopecia totalis (AT): loss of all or nearly all scalp hair;
* Alopecia universalis (AU): loss of all or nearly all scalp, face, and body hair Traditionally, a range of medications, including corticosteroids, immunotherapy, and minoxidil, are used to treat AA. However, few of these mainstay therapies are supported by robust clinical evidence, limiting the development of widely accepted clinical practice guidelines (Asfour et al., 2023). As a result of suboptimal effectiveness of traditional therapies, patients with AA, particularly those with extensive hair loss, have a persistent unmet medical need. Furthermore, the potential effects of AA on other subgroups, including patients with skin of color, remain undefined. As these subgroups have been historically underrepresented in clinical trials, an additional unmet medical need and evidence gap exists for these patients.

Recent clinical studies have demonstrated efficacy of novel treatments for AA, including ritlecitinib, a JAK3/TEC family kinase inhibitor developed and marketed by Pfizer (King et al., 2023). Ritlecitinib was approved by the US Food and Drug Administration (FDA) in June 2023 for the treatment of severe AA in adults and adolescents aged 12 years or older. Extensive information from clinical trials exists on the safety and efficacy of ritlecitinib, which, along with JAK inhibitors such as baricitinib and deuruxolitinib that are FDA approved for severe alopecia areas in adults 18 and over, have presented needed new therapeutic options for these patients. However, little is known about the clinical effectiveness of ritlecitinib in real-world clinical practice.

The objective of the current study is to evaluate patient characteristics, treatment patterns and related clinical outcomes of patients who initiated ritlecitinib to treat severe AA.

ELIGIBILITY:
Inclusion criteria:

1. Confirmed diagnosis of severe AA (as determined by the treating physician)
2. Initiated ritlecitinib for severe AA between 01 July 2023 and 28 February 2025
3. At least 12 years of age at ritlecitinib initiation
4. Has at least one additional follow-up visit/consultation after ritlecitinib initiation in which scalp hair loss was assessed
5. Has a complete medical record regarding management or treatment of AA, covering the period initial AA diagnosis until their most recent follow-up/consultation

Exclusion criteria:

1. Ever diagnosed with other types of alopecia (i.e., e.g., chemotherapy-induced alopecia, androgenic alopecia [i.e., male pattern baldness], cicatricial alopecia [i.e., scarring alopecia], postpartum alopecia, or traction alopecia), other diseases (besides AA) that can cause hair loss, or other diseases that could interfere with assessment of hair loss/regrowth
2. No documentation in the medical record of percent of scalp hair loss
3. Participated in any clinical trial involving treatment with ritlecitinib, baricitinib, deuruxolitinib, delgocitinib, brepocitinib, or upadacitinib

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients with severe AA who initiated ritlecitinib (for treatment of severe AA) at least 6 months before the start of data collection. The study assumes that treatment with ritlecitinib was per label, as indicated for severe AA among patients at least 12 years of age. Data collection will be led by physicians (or their designated clinical assistants and staff, including nurse practitioners and physician assistants) recruited to the study who specialize in dermatology and are experienced in managing patients with AA.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient demographics characteristics: race | Baseline
  Number of percentages of patients by race
Patient demographics characteristics: sex, age at initial AA diagnosis, geographic location of patient's treating dermatologist, insurance type | "Baseline" or "Day 1"
  Number of percentages of patients by sex
Patient demographics characteristics: age at initial AA diagnosis | "Baseline" or "Day 1"
  Number of percentages of patients by age at initial AA diagnosis
Patient demographics characteristics: geographic location of patient's treating dermatologist | "Baseline" or "Day 1"
  Number of percentages of patients by geographic location of patient's treating dermatologist
Patient demographics characteristics: insurance type | "Baseline" or "Day 1"
  Number of percentages of patients by insurance type
Patient clinical characteristics at initial AA diagnosis: AA disease activity | "Baseline" or "Day 1"
  Number of percentages of Patient clinical characteristics at initial AA diagnosis: AA disease activity
Patient clinical characteristics at initial AA diagnosis: SALT score | "Baseline" or "Day 1"
  Number of percentages of Patient clinical characteristics at initial AA diagnosis: SALT score
Patient clinical characteristics at initial AA diagnosis: dermatology life quality index (DLQI) score | "Baseline" or "Day 1"
  Number of percentages of Patient clinical characteristics at initial AA diagnosis: dermatology life quality index (DLQI) score
Patient clinical characteristics at initial AA diagnosis: eyebrow involvement | "Baseline" or "Day 1"
  Number of percentages of Patient clinical characteristics at initial AA diagnosis: eyebrow involvement
Patient clinical characteristics at initial AA diagnosis: eyelash involvement | "Baseline" or "Day 1"
  Number of percentages of Patient clinical characteristics at initial AA diagnosis: eyelash involvement
Patient clinical characteristics at initial AA diagnosis: beard involvement | "Baseline" or "Day 1"
  Number of percentages of Patient clinical characteristics at initial AA diagnosis: beard involvement
Patient clinical characteristics at initial AA diagnosis: AA involvement at other body locations | "Baseline" or "Day 1"
  Number of percentages of Patient clinical characteristics at initial AA diagnosis: AA involvement at other body locations
Patient treatment history: Additional treatment classes received during ritlecitinib treatment, additional treatment classes received after discontinuation of ritlecitinib, duration of each treatment class | "Day 1 through study completion, a minimum of 6-months follow-up"
Characteristics of ritlecitinib treatment: Total duration of ritlecitinib exposure, reasons for ritlecitinib discontinuation (if ritlecitinib treatment stopped before last known clinic visit), | "Day 1 through study completion, a minimum of 6-months follow-up"
Real-world clinical outcomes of ritlecitinib treatment: AA disease activity | "Day 1 through study completion, a minimum of 6-months follow-up"
  AA disease activity reported as active hair loss or inactive hair loss
Real-world clinical outcomes of ritlecitinib treatment: SALT score overall change from baseline | "Day 1 through study completion, a minimum of 6-months follow-up"
  SALT score overall change from baseline (i.e., to last observed clinic visit), as well as change from baseline to predefined post-index time points (6-, 12-, 18-, and 24-months post-index, or other relevant timepoints based on actual distribution of data). Numeric and Categorical Data: no reduction from baseline, >0%-≤25% SALT reduction, >25%-≤50% SALT reduction, >50%-≤75% SALT reduction, >75% SALT reduction; Yes/No indicator for ≥30% SALT reduction; other categories/thresholds may also be applied.
Real-world clinical outcomes of ritlecitinib treatment: SALT score | "Day 1 through study completion, a minimum of 6-months follow-up"
  Numeric data, with categorical values of <50. 50-75, 75-100, and additional categories for ≥50 (to define severe AA) and 95-100 (to defined very severe AA); alternative categories may also be applied.
Real-world clinical outcomes of ritlecitinib treatment: landmark probabilities of achieving SALT ≤20 and ≤10 | "Day 1 through study completion, a minimum of 6-months follow-up"
  Landmark probabilities of achieving SALT≤20 and SALT≤10 at 6-, 12-, 18-, and 24-months post-index date, or other relevant timepoints based on actual distribution of data.
Real-world clinical outcomes of ritlecitinib treatment: landmark probabilities of achieving a sustained SALT response | "Day 1 through study completion, a minimum of 6-months follow-up"
  Landmark probabilities of achieving a sustained SALT response at 6-, 12-, 18-, and 24-months post-index date, or other relevant timepoints based on actual distribution of data
Real-world clinical outcomes of ritlecitinib treatment: landmark probabilities of achieving ≥30% SALT score reduction from baseline at 6-, 12-, 18-, and 24-months post-index date | "Day 1 through study completion, a minimum of 6-months follow-up"
Real-world clinical outcomes of ritlecitinib treatment: beard involvement | "Day 1 through study completion, a minimum of 6-months follow-up"
  Categorical; none; minimal bear hair loss; moderate beard hair loss; severe beard hair loss; very severe or complete beard hair loss
Real-world clinical outcomes of ritlecitinib treatment: eyebrow and eyelash involvement | "Day 1 through study completion, a minimum of 6-months follow-up"
  Categorical data with values of 0 (no involvement), 1 (minimal gaps), 2 (significant gaps), or 3 (complete loss)
Real-world clinical outcomes of ritlecitinib treatment: AA involvement at other body locations | "Day 1 through study completion, a minimum of 6-months follow-up"
  Yes/no indicator for involvement at each of the following body sites: Extremities (arms, hands, legs, feet); Torso (chest, back, stomach); Pubic areas; Nasal hair; Nails
Real-world clinical outcomes of ritlecitinib treatment: DLQI score | "Day 1 through study completion, a minimum of 6-months follow-up"
Real-world clinical outcomes of ritlecitinib treatment: Patient report of feeling embarrassed or self-conscious because of AA | "Day 1 through study completion, a minimum of 6-months follow-up"
  Yes; no; as documented by the physician at each clinic visit in the post-index date period
Real-world clinical outcomes of ritlecitinib treatment: DLQI score overall change from baseline | "Day 1 through study completion, a minimum of 6-months follow-up"
Real-world clinical outcomes of ritlecitinib treatment: patient report of AA affecting social or leisure activities | "Day 1 through study completion, a minimum of 6-months follow-up"
  Yes; no; as documented by the physician at each clinic visit in the post-index date period
Real-world clinical outcomes of ritlecitinib treatment: mental health comorbidities present at last known clinic visit | "Day 1 through study completion, a minimum of 6-months follow-up"
  Yes; No; indicators for presence of specific psychiatric disorders examined in a prior systematic literature review by Lee et al. (2019)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981121